CLINICAL TRIAL: NCT02648009
Title: Metabolic Imaging of the Heart Using Hyperpolarized (13C) Pyruvate Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 332-2014
Record Dates: First submitted 2015-12-03; First posted 2016-01-06 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy | interventions — Pyruvic Acid; Injections; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Other): Arm 1
  * Group 1A: control male volunteers between 19 and 50 years of age.
  * Group 1B: control female volunteers between 19 and 50 years of age.
  * Group 1C: control male or female volunteers between 19 and 50 years of age, with the MRI scan performed twice
  * Group 1D: control male volunteers between 19 and 50 years of age.
  * Group 1E: control female volunteers between 19 and 50 years of age.
  * Group 1F: control male or female volunteers between 19 and 50 years of age, with the MRI scan performed twice
  Interventions: Drug: Hyperpolarized (13) Pyruvate Injection
- Hypertension Hypertrophy Volunteers (Other): Arm 2
  * Group 2A: patients aged 30 to 75 with hypertension and hypertrophy
  * Group 2B: patients aged 30 to 75 with non-obstructive hypertrophic cardiomyopathy (HCM).
  * Group 2C: stable outpatients with NYHA class 1-3 heart failure who have evidence of elevated LV mass (LVH), irrespective of LVEF.
  * Group 2D: stable patients with type 2 DM who have a HcA1c between 6.5-9% on oral hypoglycemic agents.
  * Group 2E: patients aged 30 to 75 with hypertrophy
  * Group 2F: patients aged 30 to 75 with hypertrophic cardiomyopathy (HCM).
  * Group 2G: stable outpatients with NYHA class 1-3 heart failure who have evidence of elevated LV mass (LVH), irrespective of LVEF.
  * Group 2H: stable patients with type 2 DM who have a HcA1c between 6.5-9% on oral hypoglycemic agents.
  Interventions: Drug: Hyperpolarized (13) Pyruvate Injection; Drug: Gadolinium

INTERVENTIONS:
Drug: Hyperpolarized (13) Pyruvate Injection — MRI with Hyperpolarized Pyruvate (13) Injection
  Other Names: Hyperpolarized Pyruvate (13) Injection
Drug: Gadolinium — MRI with Gadolinium
  Arms: Hypertension Hypertrophy Volunteers

SUMMARY:
The prevalence of congestive heart failure (CHF) in Canada is high, representing one of the health care system's most expensive diagnoses. Despite major advances in medicine, the mortality and morbidity from CHF remains great. Currently, magnetic resonance imaging (MRI) is used for non-invasive imaging of the cardiovascular system to enable the structure and anatomy of the organ to be visualized. However, current MRI methods have limitations when assessing and aiding in the management of CHF. A new imaging method has recently been developed that is showing great promise as a tool in the management of patients with CHF. Rapid imaging of biochemical reactions within myocytes using MRI has recently become possible through the use of the Dynamic Nuclear Polarization (DNP) and dissolution method. DNP-dissolution results in an intravenous contrast agent that is "hyperpolarized", producing a magnetic signal that is enhanced by up to 100,000 fold. The particular agent is carbon-13 labelled pyruvate. In this study, we demonstrate the first 13C-metabolic images of the human heart, along with the required hardware and data acquisition methods.

DETAILED DESCRIPTION:
For this study, the heart of control subjects and those with hypertension or hypertrophy will be imaged using Hyperpolarized Pyruvate 13C Injection. Different forms of Hyperpolarized Pyruvate 13C Injection are available, with the 13C labelling at different positions within the molecule. These are equivalent from a safety perspective and covered by the same Investigators Brochure, but offer different metabolic information. Two different labelling patterns are investigated in this study. If images are successfully obtained, then insights into heart failure treatments that normalize the detrimental metabolic changes may enable earlier treatment and slow disease progression to CHF, ultimately reducing the high rates of morbidity and mortality associated with this disease.

Prior to enrollment, all participants will be screened in order to ensure they meet the study's inclusion and exclusion criteria and MRI eligibility. On the day of their scan, each participant will have an intravenous line inserted and receive a glucose drink, prior to scanning. The reason for this glucose drink is that a fed versus fasted state has been found to give markedly different measurements in animal models and a choice of meal would be a source of variability. The metabolic imaging will occur shortly after this drink.

For each scan, a 1.47 g sample of [1-13C]-pyruvic acid will be hyperpolarized using a SpinLab polarizer (General Electric Co.). The solid-state sample will be dissolved to a concentration of 250 mM pyruvate at biological pH. A 0.1 mmol/kg dose (approximately 20 mL) of this solution will be injected through an intravenous line, followed by a 25 mL saline flush. The 13C image acquisition will begin at the end of the injection and will record data during every heartbeat within the single breath-hold.

Heart rate and blood pressure will be monitored non-invasively, prior to the participant being positioned within the MR scanner. Heart rate will continue to be monitored during and after the scan and the participant will be monitored by the Study's Qualified Investigator or medical designate for up to 1 hour post injection.

The 13C imaging will be preceded by the standard cardiovascular MRI workup including breath-hold cine imaging to measure ejection fraction and LV mass (~30 minutes of scan time).

Each participant in group 2 will also receive an injection of gadolinium as part of their MRI to determine evidence of late gadolinium enhancement. The recommended adult dose of 0.1ml/kg will be given. Multi-slice T1 weighted gradient echo images will be acquired. Gadolinium will be used to examine the metabolic profile in regions of scar and normal myocardium profile. LGE imaging will be performed to identify regions of scar tissue or fibrosis.

All clinical procedures will be completed under the supervision of the Qualified Investigator, or medical designate.

Each participant will receive a follow up telephone call on the 7th day following the procedure to ascertain if any study related adverse events have occurred. The length of this study for participants is a single visit that will require approximately 3 hours of their time, except for participants in Groups 1C and 1F for whom the length for the study is two visits separated by at least 2 weeks, each requiring 3 hours. The entire study is expected to take about 3 years and the results should be known approximately six months after study completion.

ELIGIBILITY:
Inclusion Criteria

* Written consent
* Age: 19 to 50 in Arm 1, 30 to 75 in Arm 2
* Group 2A and 2E participants have left-ventricular hypertrophy
* Group 2B and 2F participants have diagnosed hypertrophic cardiomyopathy
* Group 2C and 2G participants are stable outpatients with NYHA class 1-3 heart failure with evidence of elevated LV mass (LVH), irrespective of LVEF.
* Group 2D and 2H participants are stable patients with type 2 DM who have a HcA1c between 6.5-9% on oral hypoglycemic agents

Exclusion Criteria

* Contraindications to MRI or MRI contrast agents
* Hemoglobin ≤ 9.0 gm/dL (only Group 2 participants)
* Glomerular filtration rate (based on MDRD Equation) < 30 ml/min/1.73m2 (only Group 2 participants)
* Any condition leading to a life expectancy <1 year
* Medically diagnosed claustrophobia
* Have received, or are scheduled to receive, another investigational medicinal product from 1 month prior to 1 month after inclusion in this study
* BMI of less than 18.5 or greater than 32
* Group 1: medically diagnosed heart disease

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-04; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Ability of the MRI machine to produce an image of the participant's heart following an injection of Hyperpolarized Pyruvate (13C) as assessed by the physician | 2 years
  To demonstrate the first 13C-metabolic images of the human heart, along with the required hardware and data acquisition methods

SECONDARY OUTCOMES:
Imaging of participant's heart with Gadolinium | 2 years
  Gadolinium will be used to examine the metabolic profile in regions of scar and normal myocardium profile. LGE imaging will be performed to identify regions of scar tissue or fibrosis. LV scar will be reported as a percentage of LV mass.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cunningham, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Cunningham CH, Lau JY, Chen AP, Geraghty BJ, Perks WJ, Roifman I, Wright GA, Connelly KA. Hyperpolarized 13C Metabolic MRI of the Human Heart: Initial Experience. Circ Res. 2016 Nov 11;119(11):1177-1182. doi: 10.1161/CIRCRESAHA.116.309769. Epub 2016 Sep 15. PMID 27635086